CLINICAL TRIAL: NCT03723889
Title: Effect of Patent Ductus Arteriosus on Splanchnic Oxygenation at Enteral Feeding Introduction in Preterm Infants
Brief Title: Patent Ductus Arteriosus and Splanchnic Oxygenation at First Feed
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, Associate Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: SO-NIRS-PDA
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Patent Ductus Arteriosus
Keywords: Near Infrared Spectroscopy; preterm infants; intestinal complications
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PDA: Evidence of patent ductus arteriosus at echocardiography evaluation before enteral feeding introduction.
- noPDA: No evidence of patent ductus arteriosus at echocardiography evaluation before enteral feeding introduction.

SUMMARY:
Patent ductus arteriosus (PDA) is common in preterm infants. In the presence of a large PDA, significant systemic to pulmonary shunting occurs, which may results in pulmonary hyperperfusion and systemic hypoperfusion. As consequence of splanchnic hypoperfusion ensuing from left-to-right PDA shunting, a possible association between hemodynamically significant PDA and adverse gastrointestinal outcomes has been reported.

An impaired blood flow velocity in superior mesenteric artery, evaluated by Doppler ultrasound, has been previously reported before and after feeds in infants with large PDA, whereas evidence on PDA effect on splanchnic tissue oxygenation, measured by Near Infrared Spectroscopy, is scarce and controversial.

This study aims to evaluate whether splanchnic oxygenation patterns in response to enteral feeding introduction in preterm infants may be affected by PDA status.

DETAILED DESCRIPTION:
Patent ductus arteriosus (PDA) is a common condition among preterm infants. In the presence of a large PDA, significant systemic to pulmonary shunting occurs, possibly resulting in pulmonary blood flow overload and systemic hypoperfusion. A possible association with hemodynamically significant PDA and the occurrence of adverse gastrointestinal outcomes has been reported as a possible consequence of mesenteric hypoperfusion ensuing from left-to-right shunt through the PDA.

Previous attempts to assess by Doppler ultrasound the effect of PDA on blood flow velocity in superior mesenteric artery (SMA BFV) showed a decreased SMA BFV before and after feedings and attenuated postprandial increases in infants with large PDA. Near-infrared spectroscopy (NIRS) provides a non-invasive measurement of regional tissue oxygen saturation and has been previously applied in neonatal settings for the monitoring of cerebral (CrSO2) or splanchnic (SrSO2) oxygen saturation. Current evidence on the effect of PDA on SrSO2 is scarce and controversial; moreover, a possible effect of PDA on SrSO2 patterns in response to enteral feeding introduction has not been evaluated yet.

This study aims to evaluate whether SrSO2 patterns in response to enteral feeding introduction in preterm infants may be affected by the ductal status. The development of intestinal complications in relation to PDA are also evaluated.

Preterm infants <32 weeks admitted to the Neonatal Intensive Care Unit (NICU) are consecutively enrolled in the study if younger than 3 days and if no enteral feeding has been administered prior to the enrollment.

Written, informed consent to participate in the study is obtained from the parents/legal guardians of each infant before introducing enteral feeding.

At the time of enteral feeding introduction, the enrolled infants undergo a continuous monitoring of CrSO2 and SrSO2 by means of INVOS 5100 oximeter. NIRS recording is performed from 30 minutes before to 3 hours after feeding administration. CrSO2 and SrSO2 are recorded every 5 seconds. Values recorded before, during and after feeding administration are clustered into 5-minute intervals and considered for statistical analysis. Splanchnic-cerebral oxygen ratio (SCOR), which derives by the ratio between SrSO2 and CrSO2 and has been previously proposed as a valid marker for gut hypoxia-ischemia, is also calculated.

As per normal routine, an echocardiographic evaluation is performed before enteral feeding introduction, in order to evaluate hemodynamics and PDA status of the infant. In relation to the PDA status, enrolled infants are divided into the following groups: PDA (echocardiographic evidence of patent ductus arteriosus at the time of first feed) and noPDA (echocardiographic evidence of closed ductus arterious at the time of first feed).

Neonatal characteristics, including gestational age, birth weight, antenatal Doppler status, and echocardiographic PDA characteristics at the introduction of enteral feeding and the occurrence of intestinal complications during hospital stay, defined as the development of feeding intolerance (enteral feeding withholding for at least 24 hours because of gastrointestinal symptoms), necrotizing enterocolitis and spontaneous intestinal perforation, are recorded in a specific case report form.

SrSO2, CrSO2 and SCOR patterns in response to first feed are evaluated and compared between PDA and noPDA infants and adjusted for possible influencing clinical variables using a multivariate model. Moreover, the rate of intestinal complications is compared between the two study groups by chi-square test. Data are analyzed using IBM SPSS Statistic version 25 (IBM Corporation, IBM Corporation Armonk, New York, United States).

ELIGIBILITY:
Inclusion Criteria:

* gestational age <32 weeks
* no enteral feeding prior to the enrollment

Exclusion Criteria:

- major congenital malformations, including congenital heart disease

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants admitted to the Neonatal Intensive Care Unit of St. Orsola-Malpighi Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Between-group SrSO2 difference after enteral feeding introduction | 3.5 hours
  Comparison of SrSO2 values in response to the first enteral feed in infants with evidence of PDA and infants with no evidence of PDA
Between-group SCOR difference after enteral feeding introduction | 3.5 hours
  Comparison of SCOR values in response to the first enteral feed in infants with evidence of PDA and infants with no evidence of PDA

REFERENCES:
- [Background] van der Laan ME, Roofthooft MT, Fries MW, Berger RM, Schat TE, van Zoonen AG, Tanis JC, Bos AF, Kooi EM. A Hemodynamically Significant Patent Ductus Arteriosus Does Not Affect Cerebral or Renal Tissue Oxygenation in Preterm Infants. Neonatology. 2016;110(2):141-7. doi: 10.1159/000445101. Epub 2016 Apr 19. PMID 27088709
- [Background] Freeman-Ladd M, Cohen JB, Carver JD, Huhta JC. The hemodynamic effects of neonatal patent ductus arteriosus shunting on superior mesenteric artery blood flow. J Perinatol. 2005 Jul;25(7):459-62. doi: 10.1038/sj.jp.7211294. PMID 15815707
- [Background] Havranek T, Rahimi M, Hall H, Armbrecht E. Feeding preterm neonates with patent ductus arteriosus (PDA): intestinal blood flow characteristics and clinical outcomes. J Matern Fetal Neonatal Med. 2015 Mar;28(5):526-30. doi: 10.3109/14767058.2014.923395. Epub 2014 May 29. PMID 24824108
- [Background] Petrova A, Bhatt M, Mehta R. Regional tissue oxygenation in preterm born infants in association with echocardiographically significant patent ductus arteriosus. J Perinatol. 2011 Jul;31(7):460-4. doi: 10.1038/jp.2010.200. Epub 2011 Jan 20. PMID 21252960
- [Background] Martini S, Corvaglia L. Splanchnic NIRS monitoring in neonatal care: rationale, current applications and future perspectives. J Perinatol. 2018 May;38(5):431-443. doi: 10.1038/s41372-018-0075-1. Epub 2018 Feb 22. PMID 29472709
- [Derived] Martini S, Corvaglia L, Aceti A, Vitali F, Faldella G, Galletti S. Effect of Patent Ductus Arteriosus on Splanchnic Oxygenation at Enteral Feeding Introduction in Very Preterm Infants. J Pediatr Gastroenterol Nutr. 2019 Oct;69(4):493-497. doi: 10.1097/MPG.0000000000002420. PMID 31211764